CLINICAL TRIAL: NCT03014414
Title: Escalating Proportion of Weight-Loss Maintainers Via Modules Prior to Weight Loss
Brief Title: Stanford Healthy Heart Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michaela Kiernan, Senior Research Scholar, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37586; R01HL128666 (NIH)
Record Dates: First submitted 2017-01-02; First posted 2017-01-09 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fun First (Experimental): If randomized to the 12-month Fun First program, participants will attend weekly interactive small-group sessions led by health coaches for 6 months, then receive monthly phone calls from coaches for 6 months. The first 6 months consists of a 2-month module promoting enjoyment of key maintenance skills before losing weight, followed by a 4-month behavioral weight-loss program.
  Interventions: Behavioral: Fun First
- Weight Watchers (Active Comparator): If randomized to the 12-month Weight Watchers program, participants are provided with study-paid access to weekly ongoing Weight Watchers meetings led by peer meeting leaders for 12 months at Weight Watchers locations convenient to participants as well as study-paid access to Weight Watchers personalized online tools. [The study and investigative team have no financial relationship with Weight Watchers].
  Interventions: Behavioral: Weight Watchers

INTERVENTIONS:
Behavioral: Fun First — Learn key enjoyable maintenance skills before losing weight
  Arms: Fun First
Behavioral: Weight Watchers — Focus on losing weight first via convenient meetings and personalized online tools
  Arms: Weight Watchers

SUMMARY:
People with elevated blood pressure are at higher risk of having a heart attack or stroke than people with lower blood pressure. Losing a modest amount of weight-such as 15 or 20 pounds-can reduce the risk of having a heart attack or stroke. However, it can often be a struggle to maintain weight loss over time.

This study examines whether two behavioral weight-management programs can help people maintain weight loss over time. In this study, 346 adults will be randomly assigned (like flipping a coin) to one of the 12-month programs and followed for 36 months (i.e., 3 years) to see how their body weight may change.

DETAILED DESCRIPTION:
This randomized trial will test the efficacy and cost-effectiveness of novel modules administered prior to weight loss that are explicitly designed to enhance enjoyment of healthy lifestyle behaviors independent of any longer-term health effects, and thus escalate the proportion of individuals sustaining ≥7% weight loss over the long-term.

Overweight/obese individuals with elevated blood pressure will be randomized to one of two 12-month weight-management interventions (Fun First or Weight Watchers) and followed for 36 months. For Aim 1 (Primary outcome), we will test whether Fun First is more efficacious than Weight Watchers using a mediator-intervention interaction model with sufficient a priori statistical power for the interaction effect as well as the intervention and mediator main effects. The posited mediator assesses participants' change in enjoyment for four key healthy lifestyle behaviors (healthy eating, physical activity, weighing and self-nurturing) via online survey from 0-2 months. The primary outcome is the proportion of participants who lose a clinically significant amount of initial body weight and maintain it during the trial (i.e., lose >=7% of their initial body weight from 0-12 months and gain <=5 lbs from 12-36 months), assessed on clinic scales during in-person visits at the research clinic. Secondary outcomes include the proportion of individuals sustaining ≥7% weight loss over the trial assessed by digital cellular scales in participants' homes and participants' change in systolic blood pressure over the trial assessed at the research clinic.

For Aim 2 (Other pre-specified outcomes), we will test whether Fun First is more cost effective than Weight Watchers using both individual-level trial data and systems science modeling for long-term, population-level hypertension and cardiovascular disease incidence, health care and disability costs, and quality-adjusted life-years over the life course.

ELIGIBILITY:
Inclusion Criteria (BMI):

* 27 <= BMI < 45 kg/m2

Inclusion Criteria (Elevated Blood Pressure):

* Systolic blood pressure between 120-159 mmHg OR diastolic blood pressure between 80-99 mmHg. Can be on >=1 antihypertensive medications if on stable dose for past 3 months
* Systolic blood pressure <120 mmHg OR diastolic blood pressure <80 mmHg, if on stable dose of >=1 antihypertensive medications for past 3 months

Exclusion Criteria (Blood Pressure):

* Elevated blood pressure: Systolic blood pressure >=160 mmHg OR diastolic blood pressure >=100 mmHg

Exclusion Criteria (Underlying medical conditions/diseases):

* Have had a heart attack, stroke, coronary heart disease, congestive heart failure, or angina
* Have had coronary artery bypass surgery or cardiac catheterization such as percutaneous transluminal coronary angioplasty (PTCA), cath or stent placement
* Have diabetes
* Have medical contraindications to regular, unsupervised physical activity
* Have moderate to severe asthma, or chronic obstructive pulmonary disorder (also called emphysema or chronic bronchitis)
* Had cancer in the past 5 years (except non-melanoma skin cancer)
* Currently under medical care for digestive issues, gastrointestinal distress, abdominal pain, or diarrhea
* Had an organ transplant

Exclusion Criteria (Medications):

* Not stable on medications over the past 3 months (e.g., cholesterol, thyroid, estrogen-hormone, psychiatric)
* Currently taking prescription pain medications (e.g., Vicodin, Oxycodone)

Exclusion Criteria (Weight and diet related):

* Have binge eating disorder or bulimic compensatory symptoms
* Currently taking medication designed to lose weight
* Have undergone weight-loss surgery (e.g., gastric bypass, lap band)
* Have lost >10 pounds in the past 6 months
* Currently in a weight-loss program (e.g., Jenny Craig)
* Currently participating in any support groups that focus on weight or eating habits (e.g., Overeaters Anonymous)
* Currently on a special diet for a serious health condition
* Not willing to discontinue a special diet (e.g., Atkins)

Exclusion Criteria (Behavioral related):

* Planning to move in the next year
* Currently pregnant or planning to be within the next year
* Participating in another research study
* No regular access to a mobile phone and Internet
* Not able to speak, read, or understand English for informed consent
* Not willing to be randomized
* Did not complete eligibility process successfully or in a timely manner
* Staff discretion or judgement
* Live within Bay Area (e.g., ~1-hour commute from Stanford research center)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who lose a clinically significant amount of initial body weight AND maintain it during the trial (i.e., Lose >=7% of their initial body weight from 0-12 months AND gain <=5 lbs from 12-36 months), assessed by clinic scales | Baseline to 36 months
  Participants will be weighed during in-person visits at the research clinic at 0, 6, 12, 24, and 36 months

SECONDARY OUTCOMES:
Proportion of participants who lose a clinically significant amount of initial body weight AND maintain it during the trial (Lose >=7% of their initial body weight from 0-12 months AND gain <=5 lbs from 12-36 months), assessed by cellular scales | Baseline to 36 months
  Participants will be asked to weigh themselves at home on study-provided digital scales at least every 3 months from 0 to 36 months. Scales transmit body weight data via cellular technology in real time
Change in systolic blood pressure from 0-36 months | Baseline to 36 months
  Participants will have their systolic blood pressure assessed during in-person visits at the research clinic at 0, 6, 12, 24, and 36 months

OTHER OUTCOMES:
Change in self-reported enjoyment of healthy lifestyle behaviors from 0-2 months | Baseline to 2 months
  Participants will rate their enjoyment of four key healthy lifestyle behaviors (healthy eating, physical activity, weighing, self-nurturing) via online survey at 0, 2, 6, 12, 24, and 36 months [Change in enjoyment from 0-2 months is the mediator in the efficacy model]
Incremental cost-effectiveness ratio (U.S. Dollars per quality-adjusted life-years) of either weight-management intervention versus no intervention | Baseline to 36 months
  Participants will self-report their work productivity, costs, and quality-of-life via online surveys [Ratio will be based on changes in productivity, costs, and quality-adjusted life-years over the life course in the simulated cost-effectiveness model, see below for three self-reported measures incorporated into model]
Change in self-reported work productivity and activity from 6-36 months | 6 to 36 months
  Participants will report their work productivity and activity using the Work Productivity and Activity Impairment Questionnaire via online survey at 6, 12, 24, and 36 months
Change in self-reported costs of participating in the weight-management interventions from 6-36 months | 6 to 36 months
  Participants will rate their costs of participating in the weight-management interventions via online survey at 6, 12, 24, and 36 months
Change in self-reported quality of life from 0-36 months | Baseline to 36 months
  Participants will rate their quality of life using the Short Form Health Survey (SF-36) via online survey at 0, 6, 12, 24, and 36 months
Change in weight in kilograms from 0-36 months, assessed by clinic scales | Baseline to 36 months
  Participants will be weighed during in-person visits at the research clinic at 0, 6, 12, 24, and 36 months
Proportion of participants who lose >=5% of their initial body weight from 0-36 months, assessed by clinic scales | Baseline to 36 months
  Participants will be weighed during in-person visits at the research clinic at 0, 6, 12, 24, and 36 months
Change in weight in kilograms from 0-36 months, assessed by cellular scales | Baseline to 36 months
  Participants will be asked to weigh themselves at home on study-provided digital scales at least every 3 months from 0 to 36 months. Scales transmit body weight data via cellular technology in real time
Proportion of participants who lose >=5% of their initial body weight from 0-36 months, assessed by cellular scales | Baseline to 36 months
  Participants will be asked to weigh themselves at home on study-provided digital scales at least every 3 months from 0 to 36 months. Scales transmit body weight data via cellular technology in real time

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Kiernan, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
After final quality control and statistical analyses are completed, final project data will be made available to individuals who submit a written data request to the Principal Investigator. This centralized data request process provides a tracking mechanism to inform other external groups about similar analysis activities.

DOCUMENTS (1):
  • Informed Consent Form (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT03014414/ICF_000.pdf